CLINICAL TRIAL: NCT01376674
Title: Changes of T-cell-immune-status During Curative Radiotherapy in Prostate Cancer
Brief Title: T-cell-immunity During Standard Radiotherapy in Localised Prostate Cancer
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Franziska Eckert, M.D., University Hospital Tuebingen
Other Study IDs: UKT_RO_01
Record Dates: First submitted 2011-06-16; First posted 2011-06-20 (Estimated); Last update posted 2013-08-16 (Estimated); Status verified 2013-08

CONDITIONS: Prostate Cancer
Keywords: localised; prostate cancer; radiotherapy; immunology
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood mononuclear cells and serum are frozen and stored.
Oversight: Data Monitoring Committee: No

SUMMARY:
Immunological effects of radiotherapy have been described before, but not evaluated in a time-dependant manner.

In order to identify a possible time frame for combination therapies, white blood cells are isolated of samples taken at different time points before during and after standard radiotherapy in patients with localised prostate cancer. The overall activity of the T-cell-system as well as tumor-specific T-cell-response are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Localised prostate cancer (node negative)
* definitive radiotherapy
* informed consent

Exclusion Criteria:

* medication including steroids or immunosuppressants

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing standard radiotherapy for localised prostate cancer at the University Hospital of Tuebingen
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2011-03

PRIMARY OUTCOMES:
T-cell-immunity in time-course | During and 3-6 months after radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Cihan Gani, M.D., Principal Investigator — University Hospital Tuebingen; Franziska Eckert, MD, Study Director — University Hospital Tuebingen
Locations (1):
- Department of Radiation Oncology, Tübingen, Germany

REFERENCES:
- [Background] Widenmeyer M, Shebzukhov Y, Haen SP, Schmidt D, Clasen S, Boss A, Kuprash DV, Nedospasov SA, Stenzl A, Aebert H, Wernet D, Stevanovic S, Pereira PL, Rammensee HG, Gouttefangeas C. Analysis of tumor antigen-specific T cells and antibodies in cancer patients treated with radiofrequency ablation. Int J Cancer. 2011 Jun 1;128(11):2653-62. doi: 10.1002/ijc.25601. Epub 2010 Oct 8. PMID 20715115
- [Derived] Hoffmann E, Paulsen F, Schaedle P, Zips D, Gani C, Rammensee HG, Gouttefangeas C, Eckert F. Radiotherapy planning parameters correlate with changes in the peripheral immune status of patients undergoing curative radiotherapy for localized prostate cancer. Cancer Immunol Immunother. 2022 Mar;71(3):541-552. doi: 10.1007/s00262-021-03002-6. Epub 2021 Jul 16. PMID 34269847
- [Derived] Eckert F, Schaedle P, Zips D, Schmid-Horch B, Rammensee HG, Gani C, Gouttefangeas C. Impact of curative radiotherapy on the immune status of patients with localized prostate cancer. Oncoimmunology. 2018 Aug 27;7(11):e1496881. doi: 10.1080/2162402X.2018.1496881. eCollection 2018. PMID 30393582